CLINICAL TRIAL: NCT00306553
Title: Safety and Immunogenicity of a Melan-A VLP Vaccine in Advanced Stage Melanoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CYT004-MelQbG10 03
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: CYT004-MelQbG10

SUMMARY:
The purpose of this study is to evaluate a specific cellular immune response in melanoma patients that have been vaccinated with a Melan-A VLP vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent.
* Able and willing to complete all protocol requirements.
* Age: 18 years and older.
* Histological confirmed stage III or IV melanoma.
* At least one confirmed detectable target lesion
* HLA-A*0201 haplotype
* Expected survival of at least 6 months.
* Full recovery from surgery.
* Able to undergo either CT scan or MRI scan for tumor assessment.
* Wash-out period of 4 weeks after chemotherapy
* All AEs form prior anticancer therapy have resolved to ≤ Grade 1.
* Sexually active males should use adequate contraception throughout the study period and 3 months thereafter.
* Females of child bearing potential should use adequate contraception throughout the study period and 3 months thereafter, that can be oral contraception or a double-barrier local contraception (intra-uterine device plus condom or spermicidal gel plus condom), and have a negative serum pregnancy test within 4 weeks prior to the first dose of the vaccine.

Exclusion Criteria:

* Pregnant or nursing.
* Use of an investigational drug within 30 days before enrolment.
* Known or suspected brain metastases.
* Current use of an immunosuppressive drug or any concomitant medication that could potentially interfere with the study drug
* Presence of significant cardiovascular, renal, pulmonary, endocrine, infectious, neurological or bone marrow function disorders
* Serum tests positive for HIV, HBV, HCV.
* Active autoimmune diseases or severe allergies.
* Current diagnosis or history of relevant and severe psychiatric disorder that compromises the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol or to complete the study.
* Abuse of alcohol or other recreational drugs.
* Previous vaccination with a Melan-A analog peptide.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Knuth, MD, Principal Investigator — Dept. of Oncology, Univerity Hospital Zuerich, CH
Locations (2):
- Switzerland (2):
  - Dept. of Dermatology, USZ, Zurich, Canton of Zurich
  - Dept. of Oncology, USZ, Zurich, Canton of Zurich